CLINICAL TRIAL: NCT05380401
Title: Metabolic Mechanisms Induced by Enteral Docosahexaenoic Acid (DHA) and Arachidonic Acid (ARA) Supplementation in Preterm Infants
Brief Title: Metabolic Mechanisms Induced by Enteral DHA and ARA Supplementation in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20220120H; 1R01HD108646 (NIH)
Record Dates: First submitted 2022-04-22; First posted 2022-05-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Premature
Keywords: infant, premature; fatty acids; nutrition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: There will be four arms of the trial encompassing the period from enrollment to 36 weeks' postmenstrual age: (a) DHA/ARA supplement throughout the duration of the protocol, "d-on"; (b) no DHA/ARA supplement throughout the duration of the protocol, "d-off"; (c) a cross-over arm of DHA/ARA supplement from enrollment to 31 6/7 weeks post-menstrual age (PMA) then no supplement from 32 to 36 weeks' PMA, "x- on/off"; and (d) a cross-over arm of no DHA/ARA supplement till 31 6/7 weeks' then long-chain polyunsaturated fatty acids (LCPUFA) supplement from 32 to 36 weeks PMA, "x-off/on".
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DHA/ARA supplement (Other): DHA/ARA supplement throughout the duration of the protocol, "d-on"
  Interventions: Dietary Supplement: Enfamil® DHA & ARA Supplement for Special Dietary Use
- No DHA/ARA supplement (No Intervention): no DHA/ARA supplement throughout the duration of the protocol, "d-off"
- DHA/ARA initially then no supplement (Other): DHA/ARA supplement from enrollment to 31 6/7 weeks post-menstrual age (PMA) then no supplement from 32 to 36 weeks' PMA, "x- on/off"
  Interventions: Dietary Supplement: Enfamil® DHA & ARA Supplement for Special Dietary Use
- No supplement initially then DHA/ARA supplement (Other): No DHA/ARA supplement till 31 6/7 weeks' then long-chain polyunsaturated fatty acids (LCPUFA) supplement from 32 to 36 weeks PMA, "x-off/on"
  Interventions: Dietary Supplement: Enfamil® DHA & ARA Supplement for Special Dietary Use

INTERVENTIONS:
Dietary Supplement: Enfamil® DHA & ARA Supplement for Special Dietary Use — Dosage: 60 mg/kg/day of DHA and 120 mg/kg/day of ARA. Route of administration: enteral tube or by oral syringe
  Other Names: DHA/ARA Supplement
  Arms: DHA/ARA initially then no supplement; DHA/ARA supplement; No supplement initially then DHA/ARA supplement

SUMMARY:
A comprehensive analysis of the impact of exogenous enteral DHA and ARA supplementation on lipid metabolism including the production of downstream derived mediators and how this impacts important biological pathways such as metabolism, inflammation, and organogenic factors.

DETAILED DESCRIPTION:
Infants will be randomized to receive the combined enteral DHA/ARA supplement within the first 48 hours after birth to 36 weeks postmenstrual age. The randomization procedure will follow a stratified permuted block scheme to fulfill two goals: (1) randomize infants into one of four arms and (2) ensure an adequate sample size within each week of gestational age. Preterm infants will be randomized using random permuted blocks within each of the 5 birth gestational age strata. When treatment assignment is open and sample size is not overtly large, a block randomization procedure with randomly chosen block sizes can maintain treatment assignment balance and reduce the potential for selection bias. This approach will also ensure that preterm infants of all eligible gestational ages at birth are approximately equally represented in each of 4 arms of the trial, thus ensuring that important comorbidities and standard of care applicable to infants of different gestational ages at birth are also approximately equally distributed across the study arms. There is no placebo for this study. There is no blinding in this study. Consent will also be obtained from the mother of the infant, as they will be asked to provide milk samples if they're breastfeeding their infant, and maternal medical history and demographical data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* born between 25 0/7 and 29 6/7 weeks of gestation
* less than 48 hours of age at first lipid dose (The cohort is defined by gestational age rather than birth weight to avoid an over-represented sample of growth-restricted infants in birth weight defined cohorts.)

Exclusion Criteria:

* serious congenital anomalies
* conditions at birth that will require surgery prior to discharge
* imminent death such that withdrawal of intensive care support is anticipated within the first 72 hours after birth

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 328 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Fatty acid levels in plasma | Baseline to 36 weeks
  Change in lipid metabolites reflected by levels in plasma
Fatty acid levels in red blood cell (RBC) membranes | Baseline to 36 weeks
  Change in fatty acid levels in RBC membranes
Change in circulating biomarker Lipoxin A4 | Baseline to 36 weeks
  Biomarker reflective of system development and function will be measured. There are no specific levels since there is no normative data in neonates.
Change in biomarker Resolvin D1 | Baseline to 36 weeks
  Biomarker reflective of system development and function will be measured. There are no specific levels since there is no normative data in neonates.
Change in biomarker Resolvin E1 | Baseline to 36 weeks
  Biomarker reflective of system development and function will be measured. There are no specific levels since there is no normative data in neonates.
Change in Protectin/Neuroprotectin | Baseline to 36 weeks
  Levels of protectin/neuroprotectin and fatty acids in the n3 and n6 pathways will be measured.

SECONDARY OUTCOMES:
Change in infant weigh | Baseline to 36 weeks
  Recorded in grams (ounces)

OTHER OUTCOMES:
Bronchopulmonary dysplasia (BDP) | Baseline to 36 weeks
  Percentage of participants with BDP
Late-onset sepsis (LOS) | Baseline to 36 weeks
  Percentage of participants with LOS
Retinopathy of prematurity (ROP) | Baseline to 36 weeks
  Percentage of participants with ROP
Necrotizing enterocolitis (NEC) | Baseline to 36 weeks
  Percentage of participants with NEC

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Blanco, MD, MSCI-TS, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (7):
- United States (7):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Weill Cornell Medicine, New York, New York
  - University Health System, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with the funding body, NIH, summary results will be shared in ClinicalTrials.gov
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared at completion of the study when data analysis has occure.